CLINICAL TRIAL: NCT04114435
Title: Pulmonary Vascular Disease and Cardiac Performance in Extreme Preterm Infants: A Prospective Cross-sectional Study
Brief Title: Pulmonary Vascular Disease and Cardiac Performance in Extreme Preterm Infants
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriel Altit, Neonatologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-5893
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Prematurity; Extreme
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Neonatal profile: Echocardiography at:
  * 7 to 10 days of chronological age
  * 35 to 37 weeks post-menstrual age (PMA = corrected age);
  * 39 to 44 weeks PMA; Term equivalent
  Interventions: Other: Echocardiography
- Infant profile ( between 4 months and 9 months): * Echocardiography
  * Ages & stages questionnaires CAT/CLAMS assessment
  Interventions: Other: Echocardiography
- Pediatric profile (36 months and 5 years): * Echocardiography
  * Ages & stages questionnaires CAT/CLAMS assessment
  * Results from 18 months PMA Bayley will be retrieved Figure 1: Premature population - Groups Recruited simultaneously
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Diagnostic test which uses ultrasound waves to make images of the heart chambers, valves and surrounding structures

SUMMARY:
Pulmonary vascular disease and cardiac performance in extreme preterm infants: A prospective cross-sectional study

DETAILED DESCRIPTION:
The principal investigator hypothesize that premature newborns have disturbed cardiac performance and increased pulmonary pressures during neonatal life and at different pediatric ages.

The principal investigator also hypothesize that premature newborns with poor cardiac performance and/or pulmonary hypertension have higher morbidities and poorer neuro-developmental outcomes.

The principal investigator also hypothesize that premature newborns with poor cardiac performance and/or pulmonary hypertension have higher morbidities and poorer neuro-developmental outcomes and that novel echocardiography techniques will detect anomalies not uncovered by conventional imaging, and that early echocardiography may identify those with later pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <29 weeks' gestational age admitted to the NICU
* All infants born at <29 weeks' gestational age followed at MCH clinic after an admission in the NICU for prematurity <29 weeks

Exclusion Criteria:

* Congenital heart disease (except an atrial (ASD) or ventricular septal defect (VSD), or a patent ductus arteriosus (PDA))
* Congenital severe lung or airway malformation (choanal atresia, trachea-esophageal fistula or congenital pulmonary airway malformation)
* Genetic disorder (Trisomy 21).

Ages: 7 Days to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Extreme premature newborns (<29 weeks)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Heart function by echocardiography | 7-10 days of chronological age
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 35-37 weeks post-menstrual age
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 39-44 weeks PMA
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 4 months PMA
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 9 months PMA
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 36 months PMA
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance
Heart function by echocardiography | 5 years chronological
  STE allows for calculation of strain (absolute deformation) of segmental areas of the heart to provide insight on cardiac performance

SECONDARY OUTCOMES:
Neuro-developmental profile | 7-10 days of chronological age
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 35-37 weeks post-menstrual age
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 39-44 weeks PMA
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 4 months PMA
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 9 months PMA
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 36 months PMA
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography
Neuro-developmental profile | 5 years chronological
  Neuro-developmental profile of these patients at individual time points and put this profile in context of their cardiac performance by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Mcgill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No